CLINICAL TRIAL: NCT01534962
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Dose-ranging Phase II Study Assessing Ranolazine in the Maintenance of Sinus Rhythm After Electrical Cardioversion in Patients With Non-permanent Atrial Fibrillation.
Brief Title: Ranolazine in Atrial Fibrillation Following An ELectricaL CardiOversion
Acronym: RAFFAELLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAF-01; 2011-002789-18 (EudraCT Number)
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Ranolazine; Arrhythmias, Cardiac; Antiarrhythmic Agents; Cardiac Electroversion; Ranexa
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Ranolazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ranolazine low dose (Experimental): Ranolazine, low dose, oral, BID
  Interventions: Drug: Ranolazine
- Ranolazine intermediate dose (Experimental): Ranolazine, intermediate dose, oral, BID
  Interventions: Drug: Ranolazine
- Ranolazin high dose (Experimental): Ranolazine, high dose, oral, BID
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo (sugar pill), oral, BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Oral administration, BID; for a maximum of 112 days.
  Other Names: Ranexa (R)
  Arms: Ranolazine low dose
Drug: Ranolazine — Oral administration, BID; for a maximum of 112 days.
  Other Names: Ranexa (R)
  Arms: Ranolazine intermediate dose
Drug: Ranolazine — Oral administration, BID; for a maximum of 112 days.
  Other Names: Ranexa (R)
  Arms: Ranolazin high dose
Drug: Placebo — Oral administration, BID; for a maximum of 112 days.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Dose-ranging Phase II study testing the efficacy and safety of 3 doses of Ranolazine (low, intermediate and high, given BID) versus placebo in maintaining sinus rhythm after successful electrical cardioversion in patients with persistent atrial fibrillation (AFib).

After successful cardioversion and subsequent randomisation, patients report trans-telephonic EGCs on a daily basis to a central core ECG facility.

Maximum treatment duration is 112 days (16 weeks).

DETAILED DESCRIPTION:
Patients with persistent AFib are screened for eligibility and undergo direct current cardioversion (DCC). If DCC is successful (defined as persistence of sinus rhythm 2 h post-DCC) patients meeting all the inclusion criteria and none of the exclusion criteria are randomly assigned to the treatment arms (Ranolazine low, intermediate, high dose or placebo, given BID).

Transtelephonic ECG devices (TT-ECG) are used for recording of AFib recurrence to be read by a Central ECG Core Laboratory. Any symptoms indicative of AFib have to be recorded by the patient in a diary.

Study Visits are held for screening (Visit 1), at DCC and randomisation (Visit 2), one week post DCC (Visit 3), after 8 weeks of treatment (Visit 4), and at end of treatment (Visit 5). A safety follow-up telephone call is held 2 weeks after end of treatment.

12-Lead ECGs are performed at every visit.

Safety evaluations include regular safety laboratory blood and urine tests, 12-lead ECGs and the continuous recording of adverse events.

A double-dummy technique is used to ensure double-blind conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years and older
* Patients with persistent AF suitable for electrical direct current cardioversion (DCC)
* A female of childbearing potential may be enrolled providing she has a negative pregnancy test at baseline and is routinely using an effective method of birth control resulting in a low failure rate until end of study
* Able to give written informed consent before any study related procedure
* Able to attend all the visits scheduled in the study

Exclusion Criteria:

* Patients with first diagnosed AF or patients with paroxysmal AF
* Patients with long-standing persistent AF or permanent AF
* Patients having known concurrent temporary secondary causes of AF such as alcohol intoxication, pulmonary embolism, hyperthyroidism, pneumonia, hypoxemia, acute pericarditis or myocarditis
* Patients having undergone atrial catheter ablation for AF
* Patients carrying a pacemaker
* Patients with electrolytes imbalances that may cause cardiac arrhythmias, e.g. potassium < 3.5 mmol/L or > 5.5 mmol/L
* Patients with any contra-indications to Ranexa according to the drug-specific product characteristics
* Patients taking class I or Class III antiarrhythmic agents within 3 days of planned randomisation
* Patients taking beta-blockers unless used on stable doses for at least 2 weeks prior to the planned randomisation. Single doses of Intravenous beta-blockers are allowed up to 10 hours from the planned randomisation
* Patients taking Dronedarone or oral Amiodarone within 2 weeks and 3 months of planned randomisation, respectively
* Patients with a history of ECG abnormalities that in the opinion of the Investigator render the subject unsuitable for the trial, including history of congenital or a family history of long QT syndrome and a QTc interval ≥500 msec at Screening
* Patients with congestive heart failure NYHA grade III and IV;
* Patients with any serious intercurrent illness (including psychiatric and neurological disorders) which, in the opinion of the Investigator, is incompatible with the protocol.
* Patients taking Metformin at a total daily dose greater than 1000 mg.
* Patients taking Simvastatin at a total daily dose greater than 20 mg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Camm, Professor, Study Chair — Head of Clinical Cardiology; St. Gerorge's University of London, United Kingdom
Locations (4):
- Universitätsmedizin Göttingen (UMG), Kardiologie und Pneumologie, Göttingen, Lower Saxony, Germany
- FONDAZIONE IRCCS, Dip. Cardiotoracovascolare (U.C.C.), Pavia, Lombardy, Italy
- Hospital Clínic i Provincial de Barcelona, Servicio de Cardiología-Sección de Arritmias, Barcelona, Catalonia, Spain
- St. George's University of London, London, Greater London, United Kingdom

REFERENCES:
- [Derived] De Ferrari GM, Maier LS, Mont L, Schwartz PJ, Simonis G, Leschke M, Gronda E, Boriani G, Darius H, Guillamon Toran L, Savelieva I, Dusi V, Marchionni N, Quintana Rendon M, Schumacher K, Tonini G, Melani L, Giannelli S, Alberto Maggi C, Camm AJ; RAFFAELLO Investigators (see Online Supplementary Appendix for List of Participating Centers and Investigators). Ranolazine in the treatment of atrial fibrillation: Results of the dose-ranging RAFFAELLO (Ranolazine in Atrial Fibrillation Following An ELectricaL CardiOversion) study. Heart Rhythm. 2015 May;12(5):872-8. doi: 10.1016/j.hrthm.2015.01.021. Epub 2015 Jan 17. PMID 25602175

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 310 patients were screened and underwent cardioversion (CV). Of these, 241 were still in sinus rhythm 2 hours post-CV and, thus, were eligible for randomization.
  Patients who experienced an atrial fibrillation (AF) recurrence could continue the study if no medical intervention was needed and otherwise had to discontinue the study.
Period: Overall Study
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Started | 67 | 60 | 58 | 56
Completed | 30 | 34 | 34 | 24
Not Completed | 37 | 26 | 24 | 32
Not completed — Randomized but did not start treatment | 2 | 0 | 0 | 1
Not completed — Discontinued at AF recurrence | 35 | 26 | 24 | 31

BASELINE CHARACTERISTICS:
Population: ITT-population (excluding 3 randomized patients who never started study drug)
Groups:
- Placebo: Placebo, oral, BID.
- Total: Total of all reporting groups
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo | Total
Number analyzed (Participants) | 65 | 60 | 58 | 55 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (11.8) | 65.5 (8.5) | 63.6 (11.3) | 65.2 (9.5) | 65.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 12 | 14 | 54
  Male | 46 | 51 | 46 | 41 | 184
Time since AF diagnosis [Mean (Standard Deviation); unit: months] | 10.5 (24.0) | 7.2 (12.9) | 15.5 (28.2) | 6.9 (13.5) | 10.0 (20.7)

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to First Documented AF Recurrence.
Description: Time to first AF recurrence reported by patient-reported TT-ECG or 12-Lead ECG at the study site, whichever occurred first.
  Patients discontinuing the study without AF were censored at the time of the last available ECG.
Time Frame: 16 weeks (112 days)
Population: Intention-to-treat-approach that analyzed all randomised patients who took at least one dose of study medication (N=238, i.e. excluding 3 randomized patients).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Number analyzed (Participants) | 65 | 60 | 58 | 55
Days | 51.0 [9.0 to NA] — The upper limit of the CI was not calculable. | NA [68.0 to NA] — The Kaplan-Meier estimate of the median was not calculable | 117.0 [17.0 to NA] — The upper limit of the CI was not calculable. | 58.0 [16.0 to NA] — The upper limit of the CI was not calculable.

2. Secondary Outcome: Number of Patients With Documented AF Recurrences
Time Frame: 16 weeks (112 days)
Population: Intention-to-Treat (N=238)
Measure: Number; unit: participants
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Number analyzed (Participants) | 65 | 60 | 58 | 55
participants | 37 | 25 | 23 | 31

3. Secondary Outcome: Time From Randomization to First Documented and Confirmed AF Recurrence
Description: A confirmed AF recurrence was defined as a documented AF recurrence which was confirmed by a consecutive ECG performed at least 1 hour after first AF documentation.
Time Frame: 16 weeks (112 days)
Population: Intention-to-Treat (N=238)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Number analyzed (Participants) | 65 | 60 | 58 | 55
Days | 73.0 [11.0 to NA] — The upper limit of the 95% CI was not calculable. | NA [NA to NA] — The Kaplan-Meier estimate of the median and the lower/upper limit of the 95% CI was not calculable. | NA [117.0 to NA] — The Kaplan-Meier estimate of the median and the upper limit of the 95% CI was not calculable. | NA [38.0 to NA] — The Kaplan-Meier estimate of the median and the upper limit of the 95% CI was not calculable.

4. Secondary Outcome: Number of Patients With Documented and Confirmed AF Recurrences
Time Frame: 16 weeks (112 days)
Population: Intention-to-Treat
Measure: Number; unit: participants
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Number analyzed (Participants) | 65 | 60 | 58 | 55
participants | 31 | 19 | 16 | 24

5. Secondary Outcome: Time From Randomization to First Documented AF Recurrence in Patients With Sinus Rhythm 48 Hours After Cardioversion
Description: Excluding patients with early relapses (within 48 hours) while the study drug, started after cardioversion, had not yet reached steady-state.
Time Frame: 16 weeks (112 days)
Population: Modified Intention-to-Treat Population (N=217) excluding 21 patients with AF relapse within 48 hours post cardioversion
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Number analyzed (Participants) | 60 | 54 | 54 | 49
Days | 56.0 [11.0 to NA] — The upper limit of the 95% CI was not calculable. | NA [98.0 to NA] — The Kaplan-Meier estimate of the median and the upper limit of the 95% CI was not calculable. | 117.0 [18.0 to NA] — The upper limit of the 95% CI was not calculable. | 78.0 [37.0 to NA] — The upper limit of the 95% CI was not calculable.

6. Secondary Outcome: Number of Patients in Sinus Rhythm 48 Hours After Cardioversion With Documented AF Recurrence
Description: Documented AF recurrences in those patients who did not experience early relapses (within 48 hours after cardioversion)
Time Frame: 16 weeks (112 days)
Population: Modified Intention-to-Treat Population (N=217) excluding 21 patients with AF relapse within 48 hours post cardioversion
Measure: Number; unit: participants
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Number analyzed (Participants) | 60 | 54 | 54 | 49
participants | 32 | 19 | 21 | 27

ADVERSE EVENTS:
Time Frame: 16 weeks (112 days)
Arm/Group | Ranolazine Low Dose | Ranolazine Intermediate Dose | Ranolazin High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 2/65 | 3/60 | 3/58 | 4/55
Other Adverse Events (participants affected / at risk) | 51/65 | 46/60 | 42/58 | 41/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine Low Dose (N=65) | Ranolazine Intermediate Dose (N=60) | Ranolazin High Dose (N=58) | Placebo (N=55)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine Low Dose (N=65) | Ranolazine Intermediate Dose (N=60) | Ranolazin High Dose (N=58) | Placebo (N=55)
Atrial Fibrillation (Cardiac disorders) | 29 (31) | 24 (33) | 23 (27) | 27 (28)
Atrial Flutter (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Palpitations (Cardiac disorders) | 9 (11) | 11 (18) | 11 (19) | 6 (7)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (2) | 4 (7) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7) | 1 (1) | 4 (7) | 0 (0)
Asthenia (General disorders) | 4 (4) | 1 (2) | 5 (5) | 2 (2)
Chest Pain (General disorders) | 8 (9) | 7 (16) | 4 (4) | 6 (6)
Fatigue (General disorders) | 11 (13) | 10 (14) | 9 (10) | 5 (5)
Blood Creatinine increased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7) | 2 (4) | 14 (20) | 7 (8)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 5 (5) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (11) | 5 (5) | 6 (6)

LIMITATIONS AND CAVEATS:
Most of the Kaplan-Meier estimates could not be calculated due to the lower than expected number of observed events and the high variability of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less